CLINICAL TRIAL: NCT01266499
Title: A Randomized Open Label Study Evaluating the Role of Oral Antibiotics in an Aim to Eradicate Carrier State of Carbapenem- Resistant Klebsiella Pneumonia (KPC).
Brief Title: A Study Evaluating the Role of Oral Antibiotics in an Aim to Eradicate Carrier State of Carbapenem- Resistant Klebsiella Pneumonia (KPC).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, rambam68, prof, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPCCTIL
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Klebsiella Pneumoniae Carbapenemase Resistant Associated Bacteremia or Pneumonia
Keywords: Klebsiella , pneumonia, carbapenem-hydrolyzing lactamase, carbapenem-resistant Klebsiella (KPC), eradication,
MeSH Terms: conditions — Pneumonia; Klebsiella Infections; Keratoconus posticus circumscriptus | interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: will receive PO Garamycin 80mg x 4/d (Active Comparator): will receive PO Garamycin 80mg x 4/d
  Interventions: Drug: PO Garamycin 80mg x 4/d
- Group 2 : will receive PO Colistin (Polymyxin E) 100mg x 4/d (Active Comparator)
  Interventions: Drug: Colistin (Polymyxin E) 100mg x 4/d
- Group 3: will receive both medications (Active Comparator)
  Interventions: Drug: both medications
- Group 4: will not receive PO treatment (Placebo Comparator)
  Interventions: Drug: will not receive PO treatment

INTERVENTIONS:
Drug: Colistin (Polymyxin E) 100mg x 4/d — Colistin (Polymyxin E) 100mg x 4/d
  Arms: Group 2 : will receive PO Colistin (Polymyxin E) 100mg x 4/d
Drug: both medications — PO Garamycin 80mg x 4/d +PO Colistin (Polymyxin E) 100mg x 4/d
  Arms: Group 3: will receive both medications
Drug: will not receive PO treatment — will not receive PO treatment - will receive plecebo treatment
  Arms: Group 4: will not receive PO treatment
Drug: PO Garamycin 80mg x 4/d — PO Garamycin 80mg x 4/d
  Arms: Group 1: will receive PO Garamycin 80mg x 4/d

SUMMARY:
Klebsiella pneumonia, inhabitant of the digestive tract, is a frequent nosocomial pathogen. It is currently the fourth most common cause of pneumonia and fifth most common cause of bacteremia in intensive care patients (1-3).

The aim of the present randomized controlled trial is to assess the efficacy of non-absorbable oral antibiotics in the eradication of the KPC carrier state.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Patient identified as a KPC carrier.
  2. Patient capable to understand and sign informed consent
  3. Age > 18
  4. Patient capable to receive oral medication

Exclusion Criteria:

* Exclusion Criteria:

  1. Patient unable to sign informed consent
  2. Age ≤ 18
  3. Pregnant/lactating female
  4. Patient not expected to survive > 2 weeks.
  5. Patient unable or not allowed to receive oral medications
  6. A known allergy to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The specific measure that will be used to determine the effect of the intervention(s): eradication rate (%). | twice a week
  - Is this outcome measure assessing a safety issue? Select: no

CONTACTS AND LOCATIONS:
Overall Officials: Tsila Zuckerman, DR, Principal Investigator — rambam mc; ILANA OREN, Dr, Principal Investigator — Site Sub Investigator; Jacob M Rowe, Prof, Principal Investigator — Site Sub-Investigator; RENATO FINKELSTEIN, Prof, Principal Investigator — Site Sub-Investigator; Norberto Krivoy, Prof, Principal Investigator — Site Sub-Investigator; HANA Shprecher, Dr, Principal Investigator — Site Sub-Investigator; Noam Benyamini, Dr, Principal Investigator — Site Sub-Investigator; Salim Hadad, Dr, Principal Investigator — Site Sub-Investigator; Ami Neuberger, Dr, Principal Investigator — Site Sub-Investigator; Eyal Braun, Dr, Principal Investigator — Site Sub-Investigator; Ayelet Raz, Dr, Principal Investigator — Site Sub-Investigator
Locations (1):
- Rambam Mc, Haifa, Israel

REFERENCES:
- [Result] 1. Center for Disease control and prevention. National Nosocomial Infections Surveillance 9NNIS0 System report, data summary from January 1992 through June 2003. Am J Infect Control 2003:31:481-98 2. Woodford N, Tierno PM Jr, Young K, Tysall L, Palepou MF, Ward E, Painter RE, Suber DF, Shungu D, Silver LL, Inglima K, Kornblum J, Livermore DM. Antimicrobial Agents Chemother. Outbreak of Klebsiella pneumonia producing a new carbapenem-hydrolyzing class a beta-lactamase, KPC-3, in a New York Medical Center.2004;48(12):4793-9. 3. Bradford PA, Bratu S, Urban C, Visalli M, Mariano N, Landman D, Rahal JJ, Brooks S, Cebular S, Quale J Emergence of carbapenem-resistant Klebsiella species possessing the class A carbapenem-hydrolyzing KPC-2 and inhibitor-resistant TEM-30 beta-lactamases in New York City. Clin Infect Dis. 2004 1;39(1):55-60.